CLINICAL TRIAL: NCT03917264
Title: The Role of Dental Hygiene Procedures in Disruption of Healthy Homeostasis in Tissues Surrounding Dental Implants - Phase I (Ancillary Study)
Brief Title: Dental Hygiene and Peri-Implant Tissues Homeostasis Ancillary Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Royalty Research Fund - University of Washington (Other)
Responsible Party: Principal Investigator, Giorgios Kotsakis, Affiliate Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: STUDY00002852A
Record Dates: First submitted 2018-05-01; First posted 2019-04-17 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Peri-Implantitis
Keywords: implant; titanium; dental
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tooth-borne treatment (Active Comparator): Titanium curettes
  Interventions: Procedure: Peri-implantitis debridement; Other: Dental hygiene procedures
- Implant-specific treatment (Experimental): Implant brush
  Interventions: Procedure: Peri-implantitis debridement; Other: Dental hygiene procedures

INTERVENTIONS:
Procedure: Peri-implantitis debridement — Mechanical cleaning of titanium implants, peri-implantitis debridement.
Other: Dental hygiene procedures — Titanium scalers and nylon brushed used for implant cleaning

SUMMARY:
Peri-implantitis is an inflammatory disease that leads to loss of jawbone around dental implants. Recent discoveries have identified increased release of Titanium (Ti) particles around implants as being associated to peri-implantitis. In this ancillary study to the Dental Hygiene and Peri-Implant Tissues Homeostasis trial the objective is to determine potential triggers of increased Ti dissolution from the implant surface and the mechanisms by which Ti dissolution products amplify peri-implant inflammation. Results from this study will determine whether there is a differential response to Ti particles across individuals, which may alter susceptibility to peri-implantitis.

ELIGIBILITY:
Inclusion Criteria:

* Is the subject ≥ 25 years of age?
* Does the subject have an implant with a probing depth ≥ 5mm, bleeding on probing, and radiographic bone loss of > 2mm?
* Is the subject committed to the study and the required follow-up visits?

Exclusion Criteria:

- Is the subject immune compromised? Is the subject diabetic? Does the subject take steroid medication? Does the subject regularly use non-steroidal anti-inflammatories? Is the subject pregnant or intending to become pregnant during the duration of the study? Has the subject had previous implantoplasty? Did the subject take any antibiotics in the last 3 months?

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
Titanium Dissolution | 12 weeks +/- 4 weeks
  The primary outcome of the clinical trial will be titanium dissolution in periimplant plaque following treatment quantified using inductively coupled mass spectrometry (ICMS)

SECONDARY OUTCOMES:
Expression of pro-inflammatory cytokines in response to titanium | baseline
  We will determine whether PBMCs from peri-implantitis persons and controls have a differential pro-inflammatory response to titanium particles.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Kotsakis, DDS, MS, Principal Investigator — UTHealth San Antonio
Locations (2):
- United States (2):
  - UTHealth San Antonio, San Antonio, Texas
  - University of Washington School of Dentistry, Seattle, Washington